CLINICAL TRIAL: NCT05313854
Title: Diagnosis and Survival Prediction of Pancreatic Cancer by Machine Learning of Image Data
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RA-2020-455
Record Dates: First submitted 2022-03-16; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Machine Learning; Radiomics; CT; MRI; Ultrasound
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective cohort study is designed to investigate the diagnostic ability and prediction accuracy of pancreatic cancer by radiomics data and clinical data.

DETAILED DESCRIPTION:
In this study, investigators aimed to investigate the diagnostic performance and prediction accuracy of pancreatic cancer by radiomics data and clinical data, which include CT scan, MRI, PET-CT, PET-MR, ultrasound, and clinical data.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of pancreatic tumor; Must have CT / MRI / ultrasound data and pathology diagnosis

Exclusion Criteria:

Have other tumors along with pancreatic tumor; Clinical information missing

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: hospitalized patients with radiology conformed pancreatic tumor
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient overall survival | up to 3 years
  Patient overall survival, from the time of diagnosis of pancreatic tumor to the death of the patient.

SECONDARY OUTCOMES:
Pathology diagnosis | intraoperative
  Pathology diagnosis of the patient, such as adenocarcinoma, pancreatic neuroendocrine tumors, intraductal Papillary Mucinous Neoplasm, et al.

OTHER OUTCOMES:
Progression-free Survival | up to 3 years
  Patient progression-free survival, the length of time during and after the treatment of the tumor, that a patient lives with the disease but it does not get worse.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Chen, Dr, Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China

REFERENCES:
- [Derived] Xu X, Qu J, Zhang Y, Qian X, Chen T, Liu Y. Development and validation of an MRI-radiomics nomogram for the prognosis of pancreatic ductal adenocarcinoma. Front Oncol. 2023 Feb 24;13:1074445. doi: 10.3389/fonc.2023.1074445. eCollection 2023. PMID 36910599